CLINICAL TRIAL: NCT00507195
Title: Post Operative Cognitive Recovery and Neuropsychological Complications After General Anesthesia. A Comparison Between Different Techniques of Anesthesia: A Multi-Center Observational Study
Brief Title: Postanesthesia Cognitive Recovery and Neuropsychologic Complications
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Other Study IDs: pinocchio
Record Dates: First submitted 2007-07-23; First posted 2007-07-26 (Estimated); Last update posted 2007-07-26 (Estimated); Status verified 2007-05

CONDITIONS: Anesthesia Recovery Period; Delirium, Dementia, Cognitive Disorders; Neurobehavioural Manifestation; Mental Competency
Keywords: Postanethesia cognitive recovery; Postoperative delirium; hypnotics; propofol; sevoflurane; desflurane; postoperative cognitive recovery
MeSH Terms: conditions — Delirium; Dementia; Cognitive Dysfunction; Emergence Delirium | interventions — Sevoflurane; Desflurane; Propofol; Midazolam

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Hypnotics: propofol, sevoflurane, desflurane,desflurane,midazolam
  Other Names: Propofol,; sevoflurane,; desflurane,; midazolam

SUMMARY:
The study proposes to analyze the difference in the rapidity of the recovery of post operative cognition immediately after extubation and 20, 40 and 60 minutes post extubation and neuropsychological complications (delirium) after 48 hours following general anesthesia using a prospective, randomized approach. Patients undergoing any type of surgery with the exception of cranial, cardiac or thoracic surgery can be enrolled in the study.

DETAILED DESCRIPTION:
The rationale for this study comparing different types of anesthetic maintenance is based on the amount of systemic metabolic breakdown and the low repartion rates within the various tissues and the very rapid elimination of desflurane in respect to the other common inhalation and intravenous anesthetics as possible factors in the rate of recovery of cognitive function and the appearance of post operative delirium. After general anesthesia with desflurane there is less residual hypnotic agent for elimination in the circulation and tissue with respect to the amount given than with propofol or sevoflurance (1-3).

Perioperative cerebral injury correlated with surgical intervention and anesthesia can result in a decline in cognitive function (4) defining the entity of post operative cognitive dysfunction (POCD).

In this study it is possible to distinguish:

* Early POCD: attributable to anesthesia
* Long-Term POCD: could be attributable to of cognition associated with advanced age rather than to procedural effects (surgery, anesthesia, or confinement to a hospital bed)

The prevalence of POCD is higher in patients with advanced age (>70) and in cases where general anesthesia is used for highly invasive surgery (orthopedic, abdominal and thoracic surgery) (5-7). A consensus does not exist regarding tests for evaluation of POCD. In this protocol we propose to use three scales concurrently that are commonly used for evaluation of cognitive function.

Regarding neuropsychological complications, the scope of this study is to evaluate the prevalence of post operative delirium with onset during the 48 hours following the end of the surgical intervention.

Delirium fundamentally consists of three basic neuropsychological disorders:

* Visual or auditory hallucination
* Spatial-temporal disorientation
* Inappropriate language

Post operative delirium entails:

* An increase in morbidity and mortality
* An increase risk of neurological damage
* Significant discomfort for the patient, families and staff (6)

Some conditions predispose patients to the onset of post operative delirium: advanced age (>70 years old), alcohol abuse, abnormalities in the pre-operative cognitive state, and electrolyte or chemical imbalance (Na, K, glucose, etc.)

Protocol

After the induction of anesthesia, carried out using routine clinical practice determined by the anesthesiologist the patient will be assigned to either the control group or the comparison group (the assignment will have been made prior to induction). The control group will receive either propofol or sevoflurance (with or without N2O at the discretion of the anesthesiologist based on clinical needs). The comparison group will be given desflurane (end tidal 5.0 - 6.0%) for maintenance of anesthesia (with or without N2O at the discretion of the anesthesiologist based on clinical needs). According to a randomized sequence patients will be assigned in a consecutive manor to the maintenance with the control technique or with desflurane.

The objective of the study is to observe if there are differences in the point of recovery of cognition, evaluated with the appropriate test in the immediate post operative period and the onset of post operative delirium (visual or auditory hallucination, spatial or temporal disorientation, or inappropriate language) within 48 hours following surgery.

Normal care should be used in the administration of benzodiazapam premedication to patients at high risk for developing post operative delirium, but their use doe not represent criteria for exclusion from the study. In addition hypotension should be avoided (maintenance of a mean blood pressure of greater than 70 mmHg) as also intraoperative hyper ventilation (avoid hypocapnia).

Every collaborator would initially enroll 10 patients (5 control group receiving propofol or sevoflurance and 5 comparison group receiving desflurane) in order to become confident with the method of the protocol and with the evaluation methods used for measuring cognitive function.

Every collaborator and those relevant to the core study will be cited in the list of coauthors. The databases consisting of the protocol data will be at the disposal of the collaborators for further scientific work.

Statistical Analysis

The diagnostic characteristics of the patients registered will be described according to categorical variables across a table of frequency. Continuous variables will be subjected to summary statistics such as average, standard deviation, median, minimum and maximum. The differences between the groups will be subjected to verification of the significance through non-parametric (Chi Square and Fisher Exact Test for the non-continuous variables and the Mann-Whitney or the Kruskall-Wallis for associations between the continuous variables. The incidence of cardiovascular or respiratory complications, nausea and/or vomiting, shivering, neurological complications and delirium will be tabulated through table of frequency.

Criteria for Enrollment

The study includes patients of any age and ASA physical status undergoing elective surgery. All patients must have a Glascow Coma Score (GCS) equal to 15 before the intervention and they must have undergone the following:

* Informed consent about anesthesia
* Preoperative evaluation including determination of ASA physical status and GCS

Laboratory testing

* Preoperative evaluation

  * Routine laboratory tests
  * Treatment and testing appropriate to the patient's condition
* ECG
* Chest x-ray

After the induction of anesthesia which can be done according to the normal routine of the individual anesthesiologist, the patient will then be assigned according to a randomized sequence to one of the two groups:

1a) Anesthesia with propofol (total intravenous anesthesia - TVA)

1b) Anesthesia with sevoflurane (with or without N2O) 2) Anesthesia with desflurane (with or without N2O)

The anesthesiologist can use other agents (oppiods, _________, antihypertensives etc.) according to the clinical need in the judgment of the anesthesiologist. The type and quantity of drugs used in the Perioperative period must be reported on the anesthesia record.

Intra operative monitoring

* ECG
* Blood pressure (invasive or non-invasive)
* SpO2
* EtCO2
* Et halogenated agent
* Urine output

Tests Before anesthetizing the patient they will be given three cognitive tests: SOMCT, RLAS and MMSE. The same tests will be followed (repeated at emergence, after 20, 40, and 60 minutes after extubation. This will permit the evaluation of the level of recovery of cognition compared to the value obtained before anesthesia with that obtained in the three successive administrations of the tests after wake-up.

The Short Orientation Memory Concentration Test (SOMCT) investigates the patient's capacity to know the current year or month or only one of the two and to repeat in numerical order the inverse sequence of the months of the year. These variables permit the assignment of a numerical score from 0 to 28 based upon the patient's cognitive function. Higher scores indicate better cognitive function (12).

The Rancho Los Amigos Scale (RLAS) is a scale utilized to quantify the behavioral and cognitive state after acute cerebral injury. Each state corresponds to one of eight levels (I - VIII). Higher scores indicate a good state of behavior and cognition.

The Mini Mental State Examination (MMSE) is a test that is usually administered to adults or the elderly who one suspects might have a memory or character disturbance (13). This test requires the use of a pencil, a watch and some sheets of paper. The maximum attainable score is 30. A compiled score of between 24 - 30 could indicate a psychological decline in cognitive function of little importance. On the other hand scores below 24 can denote cognitive disturbance much more severe as the score decreases.

The Wake-up The start of the study period coincides with the suspension of the hypnotics (propofol/sevoflurane or desflurane). At this moment the timing of extubation begins which is at the discretion of the anesthesiologists who would evaluate the patient as usual for extubation criteria (respiratory dynamics, ability to maintain SpO2 >95%, Et CO2 between 30 - 40 mmHg, muscle strength, the presence of laryngeal reflexes, and swallowing, etc.) At that point the anesthesiologist will bring the flow of fresh gas to a value greater than that of the minute ventilation and change the circuit to an open system. The time between the suspension of anesthesia and extubation will be recorded on the patient's anesthetic record.

In order to evaluate memory quickly at termination of the anesthetic (after extubation) it would be necessary to inform the patient of the correct time and day in the immediate wake up period.

The patient is evaluated according to the Aldrete score (11) 5 minutes after the extubation ane every 5 minutes after until an Aldrete score of 9-10 is obtrained. The patient that reaches a score of 9-10 (capacity to move their extremities spontaneously and under command, to breath and cough, have a mean blood pressure between 20% of the preoperative level, to arouse themselves and the capacity to maintain an SpO2 greater than 90%) can begin to undergo cognitive testing.

At the same time interval of evaluation of the recovery of cognition, the patient will be evaluated (and treated?) for pain through use of an analogue visual scale (VAS 0 = no pain, 10 = maximum pain imaginable). The patient will then be asked for the information furnished at awakening.

During the same period the blood pressure, heart rate, ECG, SpO2 will be measured to evaluate cardiovascular, respiratory function, and the patient evaluated for nausea/vomiting, shivering and any neurological abnormalities. Episodes of hypotension (mean blood pressure less than 50 mmHg for a period greater than 5 minutes), hypertension (meant blood pressure greater than 100 mmHg for a period greater than 5 minutes) will be recorded and treated if necessary.

At 24 and 48 hours the presence of delirium will be evaluated, and in particular the appearance of alteration of spatial or temporal orientation, auditory or visual hallucinations or any inappropriate language, will be noted.

Information compiled for Patient Records

General Data This section has the aim to identify the researcher and to classify the patient. Information will be obtained regarding the patients age, sex, height and weight and the name of the medical center and the date of the intervention.

Preoperative data Needed therapy and medical condition including cardiac, respiratory, neurologic and metabolic problems prior to surgery will be recorded.

Intra-operative data This data records factors related to the intervention including anesthetic techniques utilized, fluid administered, duration of anesthesia and surgery, type of surgery and the patient's position. It is of great importance to report episodes of hypertension (systolic blood pressure <90 mmHg ) or hypertension (diastolic pressure >100 mmHg) that is protracted (duration longer than 5 minutes).

Post operative data This is data that relates to the wake up of the patients based on the three groups studied. The evaluation at wake-up and the results from the Aldrete score, the SOMCT, RLAS, and the MMSE according to the order specified in the discription of the protocol. It is important to indicated episodes of protracted hypo or hypertension and episodes of hypoxia (SpO2 < 95%) as well as the intensity of pain using the VAS (and treatment?).

ELIGIBILITY:
Inclusion Criteria:

* Adult age patients undergoing general anesthesia

Exclusion Criteria:

* Cerebral and cardiac surgery
* Surgical procedures required postoperative delayed extubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: Federico Bilotta, MD, PhD, Study Chair — University of Roma La Sapienza
Locations (1):
- Azienda Policlinico Umberto I, University of Rome La Sapienza,, Rome, Italy

REFERENCES:
- [Derived] Bilotta F, Doronzio A, Stazi E, Titi L, Zeppa IO, Cianchi A, Rosa G, Paoloni FP, Bergese S, Asouhidou I, Ioannou P, Abramowicz AE, Spinelli A, Delphin E, Ayrian E, Zelman V, Lumb P. Early postoperative cognitive dysfunction and postoperative delirium after anaesthesia with various hypnotics: study protocol for a randomised controlled trial--the PINOCCHIO trial. Trials. 2011 Jul 6;12:170. doi: 10.1186/1745-6215-12-170. PMID 21733178